CLINICAL TRIAL: NCT06893640
Title: Comparative Analysis of Cell Population Data in Chronic Lymphproliferative Disorder and Viral Disease
Brief Title: Cell Population Data in CLPD and Viral Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Randa habeeb, residant doctor, Assiut University
Other Study IDs: Cpd in CLPD and viral disease
Record Dates: First submitted 2025-03-17; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Chronic Lymphoproliferative Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group 1: Lymphoproliferative Disease
- Group 2: Viral hepatitis infection
- Group 3: Healthy control

SUMMARY:
Hematological malignancies typically arise from two major blood cell lineages: lymphoid and myeloid cells . Hematological malignancies are the fourth most frequently diagnosed cancer around the world .

Chronic lymphoproliferative disorders (CLPD) comprise a heterogeneous group of diseases characterized by uncontrolled production of lymphocytes that cause monoclonal lymphocytosis, lymphadenopathy and bone marrow infiltration. These diseases often occur in immuno-compromised individuals. There are two subsets of lymphocytes: T and B cells that regenerate uncontrollably to produce immunoproliferative disorders, which are prone to immunodeficiency, a dysfunctional immune system, and lymphocyte dysregulation. Several gene mutations have been described as causes of CLPD that can be iatrogenic or acquired .

Viral infections induce lymphocyte activation, undifferentiated lymphocyte proliferation, and antibody or cytokine/lymphokine secretion. The immune defense against viral infection is more dependent on T cells and less dependent on antibodies. Cytotoxic T cells are important in killing virally infected cells. A number of cytokines, including interferon gamma and tumor necrosis factor (TNF), are secreted by the cytotoxic T cells.1It is conceivable that the activated lymphocytes may undergo not only morphologic changes, such as an increase in size, but also alterations in cytoplasmic composition as compared to their normal 'resting' counterparts .

Beyond the differential leukocyte count, modern hematological analyzers provide additional quantitative data known as "cell population data (CPD) which is regarded as the fingerprint of a blood cell at a given moment. CPD parameters harbor information associated with cell morphology and offer detailed information about the size, complexity, and fluorescence characteristics of different cell populations, potentially aiding in the diagnosis and management of various haematological conditions .

There has been no comprehensive study on the usefulness of cell population data (CPD) parameters as a screening tool in the discrimination of non-neoplastic(viral infection) and neoplastic haematological disorders such CLPD.

the aim of the study evalute clinical utility of CPD parameters generated by haematological analyser in diagnosis of both CLPD &viral infection 2-to compare performance of CPD parameters with other established diagnostic &prognostic markers in CLPD

ELIGIBILITY:
Inclusion Criteria:

* 1-Age > 18 years old 2- Patient newly diagnosed CLPD according to the recent WHO classification; based on bone marrow examination, immunophenotyping &/or LN biopsy 3- Patients are newly diagnosed with viral hepatitis infection based on viral serology

Exclusion Criteria:

* 1- patient on treatment 2- Patient has both chronic lymphoproliferative disorders and viral hepatitis infection 3- Patient has any other' hematological disease 4- Patient has any chronic disease affect hematological parameters. 5- patient with incomplete medical records

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Lymphoproliferative Disease: 59 patients
  * Viral hepatitis infection: 59 patients
  * Healthy control : 59
Sampling Method: Non-Probability Sample
Enrollment: 177 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Leukocyte cell population data | baseline
  Leukocyte cell population data (CPD)